CLINICAL TRIAL: NCT06019221
Title: Pediatric Relapsing Polychondritis : Diagnosis and Management in a French Retrospective Study
Acronym: PRP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8783
Record Dates: First submitted 2023-08-24; First posted 2023-08-31 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-08

CONDITIONS: Relapsing Polychondritis
Keywords: Polychondritis; Relapsing Polychondritis; Pediatric Relapsing Polychondritis
MeSH Terms: conditions — Polychondritis, Relapsing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The incidence in pediatrics is very low (about 3.5 per million per year according to a 2015 study) and therefore the data on the pathology very poor, especially on the therapeutic level.

Without appropriate treatment, the disabling sequelae, even involving the vital prognosis, are significant. However, in paediatrics, therapeutic habits have been extrapolated from adult data and lack precision.

Existing treatments are almost composed of immunomodulatory and/or immunosuppressive treatments. Different therapeutic lines have been introduced over the years and a better understanding of the pathology. More recently, biotherapies have been introduced in this pathology, but data on their effectiveness remain limited. Data on the evolution under therapy in children are thus still poor.

Complications related to the pathology that can jeopardize the vital prognosis and the response to treatment for this pathology deserve to be studied in order to be known and if possible avoided.

The aim of the study is to describe French practices and compare the lines of treatment proposed for juvenile atrophic polychondritis.

ELIGIBILITY:
Inclusion criteria:

* Minor subject aged 1 to 17 years
* Diagnosis of atrophic polychondritis between 01/01/2008 to 31/12/2022.
* Subject (and/or his parental authority) who has not expressed, after being informed, his opposition to the reuse of his data for the purposes of this research.

Exclusion criteria:

* Subject (or his parents) having expressed his (their) opposition to participating in the study
* Associated pathologies that cannot be related to the diagnosis of atrophic polychondritis and whose prognosis can lead to biases in the efficacy and/or complications related to treatments.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Minor subject aged 1 to 17 years having atrophic polychondritis
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-02-18 (Actual); Primary Completion 2024-01-18 (Estimated); Study Completion 2024-01-18 (Estimated)

PRIMARY OUTCOMES:
Therapeutic effectiveness of the various treatments proposed depending on the degree of initial clinical involvement | Files analysed retrospectively from from January 01, 2008 to December 31, 2022 will be examined
  The aim of this study is to bring together the experiences of the various reference and competence centers in France concerning the clinical presentation, management and follow-up of children with relapsing polychondritis.

CONTACTS AND LOCATIONS:
Overall Officials: Ariane ZALOSZYC, MD, Study Director — University Hospitals of Strasbourg
Locations (1):
- Service de Pédiatrie 1 - CHU de Strasbourg - France, Strasbourg, France